CLINICAL TRIAL: NCT06571630
Title: Polish Mother's Memorial Hospital Research Institute - Familial Hypercholesterolemia Registry
Brief Title: PMMHRI - Familial Hypercholesterolemia Registry
Acronym: FH-Registry
Status: Recruiting | Type: Observational
Sponsor: Polish Mother Memorial Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PMMHRI-FH-Registry
Record Dates: First submitted 2024-08-08; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Familial Hypercholesterolemia
Keywords: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The registry is maintained at the Regional Centre for Rare Diseases, established in 2016, within Polish Mother's Memorial Hospital Research Institute. This facility diagnoses and treats over 80 distinct rare diseases in patients from across the country, including those with phenotypically or genetically confirmed familial hypercholesterolemia (FH).

DETAILED DESCRIPTION:
All consecutive patients diagnosed with FH, including both children and adults, are being enrolled from December 2018 to May 2024. Each patient receives a consultation with a clinical geneticist and a dietitian, who provide recommendations for cascade screening among family members and promote a healthy and balanced diet. The study includes all index cases, with children also serving as index cases.

The PMMHRI FH registry is managed by physicians from the RCRD, who exclusively make all diagnostic and treatment decisions. The purpose of the registry is to investigate the clinical characteristics, diagnosis, management, achievement of therapeutic goals, and outcomes of FH patients. Inclusion criteria are based on phenotypic or genetic diagnosis of FH. Phenotypic diagnosis is conducted using the Dutch Lipid Clinic Network criteria for adults, and the Simon Broome criteria for children. During the baseline visit, comprehensive data collection includes all available lipidogram results, aiming to obtain naive LDL-C values, highest values, and treated values. All data collected during the enrollment period are included in the study.

ELIGIBILITY:
Inclusion Criteria:

* FH diagnosis

Exclusion Criteria:

-

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients diagnosed with FH, including both children and adults,
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Therapeutic goals achivement | 5 years
  For each patient, we collect data on the levels of all lipid profile fractions: such as total cholesterol [mg/dl], low density lipoprotein cholesterol - LDL [mg/dl], high density lipoprotein cholesterol HDL [mg/dl], triglycerides [mg/dl], non-HDL [mg/dl] and lipoprotein(a) during both dual and triple therapy. Additionally, we will assess the achievement of the therapeutic target as defined by the ESC guidelines. The therapeutic target for each patient will be evaluated individually based on their risk, in accordance with the ESC guidelines.

CONTACTS AND LOCATIONS:
Locations (1):
- Polish Mother Memorial Research Institute (PMMHRI) in Lodz, Poland, Lodz, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lewek J, Konopka A, Starostecka E, Penson PE, Maciejewski M, Banach M. Clinical Features of Familial Hypercholesterolemia in Children and Adults in EAS-FHSC Regional Center for Rare Diseases in Poland. J Clin Med. 2021 Sep 22;10(19):4302. doi: 10.3390/jcm10194302. PMID 34640319
- [Background] European Atherosclerosis Society Familial Hypercholesterolaemia Studies Collaboration. Familial hypercholesterolaemia in children and adolescents from 48 countries: a cross-sectional study. Lancet. 2024 Jan 6;403(10421):55-66. doi: 10.1016/S0140-6736(23)01842-1. Epub 2023 Dec 12. PMID 38101429
- [Background] EAS Familial Hypercholesterolaemia Studies Collaboration (FHSC). Global perspective of familial hypercholesterolaemia: a cross-sectional study from the EAS Familial Hypercholesterolaemia Studies Collaboration (FHSC). Lancet. 2021 Nov 6;398(10312):1713-1725. doi: 10.1016/S0140-6736(21)01122-3. Epub 2021 Sep 7. PMID 34506743